CLINICAL TRIAL: NCT02711007
Title: A Phase II Trial of Apatinib in Relapsed and Unresectable High-grade Osteosarcoma After Failure of Standard Multimodal Therapy
Brief Title: Apatinib for Advanced Osteosarcoma After Failure of Standard Multimodal Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: GUO WEI (Other)
Responsible Party: Sponsor-Investigator, GUO WEI, The Director of the Musculoskeletal Tumor Center of Peking University People's Hospital and the Principal Investigator of this study, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma
Record Dates: First submitted 2016-03-13; First posted 2016-03-17 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Osteosarcoma; Metastasis
Keywords: osteosarcoma; metastasis; advanced; apatinib
MeSH Terms: conditions — Osteosarcoma; Neoplasm Metastasis | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- apatinib (Experimental): apatinib 750mg tablet or 500mg tablet by mouth, Qd half an hour after dinner
  Interventions: Drug: apatinib

INTERVENTIONS:
Drug: apatinib — Apatinib is a small-molecule VEGFR tyrosine kinase inhibitor, similar to vatalanib (PTK787), but with a binding affinity 10 times that of vatalanib or sorafenib.

SUMMARY:
After standard multimodal therapy, the prognosis of relapsed and unresectable high-grade osteosarcoma is dismal and unchanged over the last decades.Thus, the investigators explored apatinib activity in patients with relapsed and unresectable osteosarcoma after the failure of first-line or second-line chemotherapy. Patients >16 years, progressing after standard treatment, were eligible to receive 500 mg or 750 mg of apatinib once daily until progression or unacceptable toxicity. The primary end point was progression-free survival (PFS) at 4 months and objective response rate (ORR). Secondary objectives were PFS, overall survival (OS), clinical benefit rate (CBR), defined as no progression at 6 months and safety.

DETAILED DESCRIPTION:
Patients

Eligible patients should have the following characteristics: age >16 years; diagnosis of high-grade osteosarcoma confirmed histologically and reviewed centrally; prior treatment (completed >4 weeks before trial entry) consisted of standard high-grade osteosarcoma chemotherapy agents including doxorubicin, cisplatin, high-dose methotrexate, and ifosfamide; metastatic relapsed and unresectable progressive disease (PD); Eastern Cooperative Oncology Group performance status 0-1 with a life expectancy >3 months; adequate renal, hepatic, and hemopoietic function. Additionally, the investigators require normal or controlled blood pressure, as well as surgery and/or radiotherapy completion at least 1 month before enrollment. All enrolled patients showed radiological evidence of disease progression and the lesion could be evaluated according to RECIST 1.1 before treatment start.

Treatment

Patients are planned to be treated with a dose of apatinib 500 mg(BSA ≤1.5) or 750mg(BSA>1.5) once daily. The dose was reduced or temporarily suspended according to predefined rules and after considering any observed toxicity, which was assessed according to the Common Terminology Criteria for Adverse Events version 3.0. Following adverse event resolution, apatinib can be restarted at the maximally tolerated dose and continued until progression, unacceptable toxicity or patient refusal. The study was approved by participating hospital review boards, and conducted according to the Declaration of Helsinki and the International Conference on Harmonization of Good Clinical Practice guidelines. Each patient provided written informed consent.

Efficacy Assessment

Before starting treatment, patients should be staged with chest and abdomen computed tomography (CT) and magnetic resonance imaging (MRI) (whenever indicated by the clinical situation). And all those patients should be tested by Immunohistochemistry of the VEGFR-2 over-expression of the paraffin embedded samples of the lesion or mRNA testing VEGFR-2 over-expression of the fresh specimen. Baseline assessment included also full blood count, serum chemistry, electrocardiogram and physical examination. In light of its potential role in osteosarcoma response assessment, [18F]2-fluoro-2-deoxy-D-glucose-positron emission tomography (FDG-PET) is suggested but not mandated for patient enrollment, and its impact on tumor response assessment was purely exploratory. All tests were repeated after 2 months and, thereafter, at 2-month intervals unless there were toxic effects or disease progression suspicion. Response was assessed by CT/MRI scan according to RECIST 1.1. Thus, both complete and partial remission needed confirmation within 4 weeks of when a response was first demonstrated. Stable disease (SD) was confirmed after a minimum of 8 weeks. The investigators thoroughly probe for and record any sign(s) of treatment-induced improvement, be it minor response (MR) as tumor shrinkage <30%, and/or nondimensional tumor responses including Hounsfield unit measured tissue density changes or osteoid matrix calcification.

The primary end point progression-free survival (PFS) at 4 months is calculated from the date of treatment start until the time of disease progression or death, whichever came first. Patients alive and free from progression would be censored. Secondary end points included the following: PFS; OS; overall response rate, defined as complete responses (CRs) + partial responses (PRs) + MRs; disease control rate (overall response rate + SDs); patterns of nondimensional response; clinical benefit rate (CBR) (PFS rate at 4 months) and duration of response. Duration of response is calculated from the day of first response assessment until either progression/death (event) or last day of follow-up (censored). Last, the investigators evaluate any clinical improvement by means of the Pain Analgesic Score via the Brief Pain Inventory (BPI) score form that was filled in by patients themselves. Analgesic medication use was recorded according to the analgesic score: 0 = none; 1 = minor analgesics; 2 = tranquillizers, antidepressants, muscle relaxants and steroids; 3 = mild narcotics; 4 = strong narcotics.

ELIGIBILITY:
Inclusion Criteria:

* age >16 years;
* diagnosis confirmed histologically and reviewed centrally;
* prior treatment (completed >4 weeks before trial entry) consisted of standard high-grade osteosarcoma chemotherapy agents including doxorubicin, cisplatin, high- dose methotrexate, and ifosfamide; metastatic relapsed and unresectable progressive disease (PD);
* Eastern Cooperative Oncology Group performance status 0-1 with a life expectancy >3 months;
* adequate renal, hepatic, and hemopoietic function;
* normal or controlled blood pressure;
* surgery and/or radiotherapy completion at least 1 month before enrollment.

Exclusion Criteria:

* no pulmonary artery or venous tumor embolus;
* previously exposed to other TKIs;
* central nervous system metastasis;
* have had other kinds of malignant tumors at the same time;
* cardiac insufficiency or arrhythmia;
* uncontrolled complications, such as diabetes mellitus and so on;
* coagulation disorders;
* urine protein≥ ++;
* pleural or peritoneal effusion that needs to be handled by surgical treatment;
* combined with other infections or wounds.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival, PFS | 4 months
  calculated from the date of treatment start until the time of disease progression or death, whichever comes first.
Objective response rate, ORR | 3 months
  CR+PR at 3 months

SECONDARY OUTCOMES:
Overall survival, OS | 12 months
  calculated from the date of treatment start until last follow-up or death, whichever comes first.
Clinical benefit rate, CBR | 6 months
  CR+PR+SD at 6 months
Duration of response, DOR | 6 months
  Duration of response is calculated from the day of first response assessment until either progression/death (event) or last day of follow-up (censored).

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, M.D. Ph.D., Study Chair — Chinese Medical Association--Sarcoma group
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
the investigator decide to share all the statistical analysis plan, clinical study report and anlytic code to other researchers

REFERENCES:
- [Background] Bernthal NM, Federman N, Eilber FR, Nelson SD, Eckardt JJ, Eilber FC, Tap WD. Long-term results (>25 years) of a randomized, prospective clinical trial evaluating chemotherapy in patients with high-grade, operable osteosarcoma. Cancer. 2012 Dec 1;118(23):5888-93. doi: 10.1002/cncr.27651. Epub 2012 May 30. PMID 22648705
- [Background] Bielack S, Jurgens H, Jundt G, Kevric M, Kuhne T, Reichardt P, Zoubek A, Werner M, Winkelmann W, Kotz R. Osteosarcoma: the COSS experience. Cancer Treat Res. 2009;152:289-308. doi: 10.1007/978-1-4419-0284-9_15. PMID 20213397
- [Background] Kempf-Bielack B, Bielack SS, Jurgens H, Branscheid D, Berdel WE, Exner GU, Gobel U, Helmke K, Jundt G, Kabisch H, Kevric M, Klingebiel T, Kotz R, Maas R, Schwarz R, Semik M, Treuner J, Zoubek A, Winkler K. Osteosarcoma relapse after combined modality therapy: an analysis of unselected patients in the Cooperative Osteosarcoma Study Group (COSS). J Clin Oncol. 2005 Jan 20;23(3):559-68. doi: 10.1200/JCO.2005.04.063. PMID 15659502
- [Background] Cheong JH, Hyung WJ, Chen J, Kim J, Choi SH, Noh SH. Surgical management and outcome of metachronous Krukenberg tumors from gastric cancer. J Surg Oncol. 2004 Jul 15;87(1):39-45. doi: 10.1002/jso.20072. PMID 15221918
- [Background] van Rijk-Zwikker GL, Nooy MA, Taminiau A, Kappetein AP, Huysmans HA. Pulmonary metastasectomy in patients with osteosarcoma. Eur J Cardiothorac Surg. 1991;5(8):406-9. doi: 10.1016/1010-7940(91)90184-l. PMID 1910847
- [Background] Thompson RC Jr, Cheng EY, Clohisy DR, Perentesis J, Manivel C, Le CT. Results of treatment for metastatic osteosarcoma with neoadjuvant chemotherapy and surgery. Clin Orthop Relat Res. 2002 Apr;(397):240-7. doi: 10.1097/00003086-200204000-00028. PMID 11953615
- [Background] Navid F, Willert JR, McCarville MB, Furman W, Watkins A, Roberts W, Daw NC. Combination of gemcitabine and docetaxel in the treatment of children and young adults with refractory bone sarcoma. Cancer. 2008 Jul 15;113(2):419-25. doi: 10.1002/cncr.23586. PMID 18484657
- [Background] Berger M, Grignani G, Ferrari S, Biasin E, Brach del Prever A, Aliberti S, Saglio F, Aglietta M, Fagioli F. Phase 2 trial of two courses of cyclophosphamide and etoposide for relapsed high-risk osteosarcoma patients. Cancer. 2009 Jul 1;115(13):2980-7. doi: 10.1002/cncr.24368. PMID 19452540
- [Background] Saylors RL 3rd, Stine KC, Sullivan J, Kepner JL, Wall DA, Bernstein ML, Harris MB, Hayashi R, Vietti TJ; Pediatric Oncology Group. Cyclophosphamide plus topotecan in children with recurrent or refractory solid tumors: a Pediatric Oncology Group phase II study. J Clin Oncol. 2001 Aug 1;19(15):3463-9. doi: 10.1200/JCO.2001.19.15.3463. PMID 11481351
- [Background] Miser JS, Kinsella TJ, Triche TJ, Tsokos M, Jarosinski P, Forquer R, Wesley R, Magrath I. Ifosfamide with mesna uroprotection and etoposide: an effective regimen in the treatment of recurrent sarcomas and other tumors of children and young adults. J Clin Oncol. 1987 Aug;5(8):1191-8. doi: 10.1200/JCO.1987.5.8.1191. PMID 3114435
- [Background] McNall-Knapp RY, Williams CN, Reeves EN, Heideman RL, Meyer WH. Extended phase I evaluation of vincristine, irinotecan, temozolomide, and antibiotic in children with refractory solid tumors. Pediatr Blood Cancer. 2010 Jul 1;54(7):909-15. doi: 10.1002/pbc.22460. PMID 20405511
- [Background] Bomgaars LR, Bernstein M, Krailo M, Kadota R, Das S, Chen Z, Adamson PC, Blaney SM. Phase II trial of irinotecan in children with refractory solid tumors: a Children's Oncology Group Study. J Clin Oncol. 2007 Oct 10;25(29):4622-7. doi: 10.1200/JCO.2007.11.6103. PMID 17925558
- [Background] Cosetti M, Wexler LH, Calleja E, Trippett T, LaQuaglia M, Huvos AG, Gerald W, Healey JH, Meyers PA, Gorlick R. Irinotecan for pediatric solid tumors: the Memorial Sloan-Kettering experience. J Pediatr Hematol Oncol. 2002 Feb;24(2):101-5. doi: 10.1097/00043426-200202000-00009. PMID 11990694
- [Background] Debiec-Rychter M, Sciot R, Le Cesne A, Schlemmer M, Hohenberger P, van Oosterom AT, Blay JY, Leyvraz S, Stul M, Casali PG, Zalcberg J, Verweij J, Van Glabbeke M, Hagemeijer A, Judson I; EORTC Soft Tissue and Bone Sarcoma Group; Italian Sarcoma Group; Australasian GastroIntestinal Trials Group. KIT mutations and dose selection for imatinib in patients with advanced gastrointestinal stromal tumours. Eur J Cancer. 2006 May;42(8):1093-103. doi: 10.1016/j.ejca.2006.01.030. Epub 2006 Apr 18. PMID 16624552
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Sleijfer S, Ray-Coquard I, Papai Z, Le Cesne A, Scurr M, Schoffski P, Collin F, Pandite L, Marreaud S, De Brauwer A, van Glabbeke M, Verweij J, Blay JY. Pazopanib, a multikinase angiogenesis inhibitor, in patients with relapsed or refractory advanced soft tissue sarcoma: a phase II study from the European organisation for research and treatment of cancer-soft tissue and bone sarcoma group (EORTC study 62043). J Clin Oncol. 2009 Jul 1;27(19):3126-32. doi: 10.1200/JCO.2008.21.3223. Epub 2009 May 18. PMID 19451427
- [Background] Linch M, Miah AB, Thway K, Judson IR, Benson C. Systemic treatment of soft-tissue sarcoma-gold standard and novel therapies. Nat Rev Clin Oncol. 2014 Apr;11(4):187-202. doi: 10.1038/nrclinonc.2014.26. Epub 2014 Mar 18. PMID 24642677
- [Background] Schoffski P, Cornillie J, Wozniak A, Li H, Hompes D. Soft tissue sarcoma: an update on systemic treatment options for patients with advanced disease. Oncol Res Treat. 2014;37(6):355-62. doi: 10.1159/000362631. Epub 2014 Apr 17. PMID 24903768
- [Background] Grignani G, Palmerini E, Dileo P, Asaftei SD, D'Ambrosio L, Pignochino Y, Mercuri M, Picci P, Fagioli F, Casali PG, Ferrari S, Aglietta M. A phase II trial of sorafenib in relapsed and unresectable high-grade osteosarcoma after failure of standard multimodal therapy: an Italian Sarcoma Group study. Ann Oncol. 2012 Feb;23(2):508-16. doi: 10.1093/annonc/mdr151. Epub 2011 Apr 28. PMID 21527590
- [Background] Yoo C, Lee J, Rha SY, Park KH, Kim TM, Kim YJ, Lee HJ, Lee KH, Ahn JH. Multicenter phase II study of everolimus in patients with metastatic or recurrent bone and soft-tissue sarcomas after failure of anthracycline and ifosfamide. Invest New Drugs. 2013 Dec;31(6):1602-8. doi: 10.1007/s10637-013-0028-7. Epub 2013 Sep 14. PMID 24037083
- [Background] Grignani G, Palmerini E, Ferraresi V, D'Ambrosio L, Bertulli R, Asaftei SD, Tamburini A, Pignochino Y, Sangiolo D, Marchesi E, Capozzi F, Biagini R, Gambarotti M, Fagioli F, Casali PG, Picci P, Ferrari S, Aglietta M; Italian Sarcoma Group. Sorafenib and everolimus for patients with unresectable high-grade osteosarcoma progressing after standard treatment: a non-randomised phase 2 clinical trial. Lancet Oncol. 2015 Jan;16(1):98-107. doi: 10.1016/S1470-2045(14)71136-2. Epub 2014 Dec 11. PMID 25498219
- [Background] Lammli J, Fan M, Rosenthal HG, Patni M, Rinehart E, Vergara G, Ablah E, Wooley PH, Lucas G, Yang SY. Expression of Vascular Endothelial Growth Factor correlates with the advance of clinical osteosarcoma. Int Orthop. 2012 Nov;36(11):2307-13. doi: 10.1007/s00264-012-1629-z. Epub 2012 Aug 2. PMID 22855059
- [Background] Li J, Qin S, Xu J, Guo W, Xiong J, Bai Y, Sun G, Yang Y, Wang L, Xu N, Cheng Y, Wang Z, Zheng L, Tao M, Zhu X, Ji D, Liu X, Yu H. Apatinib for chemotherapy-refractory advanced metastatic gastric cancer: results from a randomized, placebo-controlled, parallel-arm, phase II trial. J Clin Oncol. 2013 Sep 10;31(26):3219-25. doi: 10.1200/JCO.2013.48.8585. Epub 2013 Aug 5. PMID 23918952
- [Background] Aras M, Erdil TY, Dane F, Gungor S, Ones T, Dede F, Inanir S, Turoglu HT. Comparison of WHO, RECIST 1.1, EORTC, and PERCIST criteria in the evaluation of treatment response in malignant solid tumors. Nucl Med Commun. 2016 Jan;37(1):9-15. doi: 10.1097/MNM.0000000000000401. PMID 26440568
- [Background] Semiglazov V. RECIST for Response (Clinical and Imaging) in Neoadjuvant Clinical Trials in Operable Breast Cancer. J Natl Cancer Inst Monogr. 2015 May;2015(51):21-3. doi: 10.1093/jncimonographs/lgv021. PMID 26063880
- [Background] Young J, Badgery-Parker T, Dobbins T, Jorgensen M, Gibbs P, Faragher I, Jones I, Currow D. Comparison of ECOG/WHO performance status and ASA score as a measure of functional status. J Pain Symptom Manage. 2015 Feb;49(2):258-64. doi: 10.1016/j.jpainsymman.2014.06.006. Epub 2014 Jul 1. PMID 24996034
- [Background] Broderick JM, Hussey J, Kennedy MJ, O' Donnell DM. Patients over 65 years are assigned lower ECOG PS scores than younger patients, although objectively measured physical activity is no different. J Geriatr Oncol. 2014 Jan;5(1):49-56. doi: 10.1016/j.jgo.2013.07.010. Epub 2013 Sep 5. PMID 24484718

DOCUMENTS (2):
  • Study Protocol (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT02711007/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT02711007/SAP_001.pdf